CLINICAL TRIAL: NCT04473365
Title: Rapid Diagnostic Profiling of SARS-CoV-2 in the Context of Persistent Immune Activation in Sub-Saharan Africa (Profile-Cov)
Brief Title: Rapid Diagnostic Profiling of SARS-CoV-2 (COVID-19)
Acronym: Profile-Cov
Status: Completed | Type: Observational
Sponsor: Mekelle University (Other)
Collaborators: Ethiopian Public Health Institute (Other Government); Liverpool School of Tropical Medicine (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Tigray Health Research Institute (Unknown)
Responsible Party: Principal Investigator, Prof. Dawit Wolday, Associate Professor of Medicine, Mekelle University
Other Study IDs: RIA2020EF-2905
Record Dates: First submitted 2020-07-11; First posted 2020-07-16 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: SARS-CoV-2; COVID-19
Keywords: Immune profile; Serology; Antibody test; Antigen test; SARS-CoV-2; COVID-19; Immune response; Severity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples and PBMC biobanking for further analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Without parasite: For secondary outcome: effect of co-infection with parasite on COVID-19 severity Group 1 will constitute those without parasite co-infection
- With parasite: For secondary outcome: effect of co-infection with parasite on COVID-19 severity Group 2 will constitute those with parasite co-infection
  Interventions: Other: Intestinal parasite

INTERVENTIONS:
Other: Intestinal parasite — Pre-existing intestinal parasite infection present or absent at time of admission
  Other Names: Without intestinal parasite
  Groups: With parasite

SUMMARY:
The investigators will evaluate the profile of the immune response of Ethiopian population and examine its relationship with the noted low CD4+ T-cell count and underlying immune activation status among participants with COVID-19 and will compare results with those residing in Europe. In addition, this project will evaluate the performance of various rapid diagnostic tests (RDTs) for SARS-CoV-2, taking into account the above-determined immune system characteristics. We will also evaluate the effect of co-infection with parasites on COVID-19 severity

DETAILED DESCRIPTION:
In December 2019, a cluster of patients with pneumonia of unknown aetiology was linked to an infection with a novel coronavirus - the SARS-CoV-2. Since then, the infection has become pandemic and spread affecting almost every country in the world. Knowledge of virus dynamics and the host's immune response to it is essential to understanding the pathogenesis as well as in formulating diagnostic, therapeutic and preventive strategies. There are no studies, however, related to these issues, particularly in Sub-Saharan Africa (SSA) context. Previous studies by the investigators have shown that the immune profile of healthy Ethiopians shows evidence of chronic immune activation with significant low naïve cells but high activated memory cells, of both CD4+ and CD8+ T-cell sub populations. The above immune system characteristics of Ethiopians as compared to Europeans led the investigators to the assumption that these could contribute to the pathogenesis of and severity of clinical presentation of COVID-19. Persistent immune activation due to continuous infections with helminths is common in the entire SSA region. Such activation usually skewes the immune system towards T helper (Th)-2-type responses. The immune response against SARS-CoV-2 is typically of so called "cytokine storm". Here, the investigators hypothesize that SARS-CoV-2 infection induced immune activation as observed in patients in the industrialized world (with concomitant cytokine storms and extensive non-specific CD8 T-cell cytotoxicity) might be more prominent than in people from SSA, due to the Th2 profile of their immune system.

The investigators propose to study the profile of the immune response of Ethiopian population and will examine its relationship with the noted low CD4+ T-cell count and underlying immune activation status among patients with COVID-19 and will compare results with those residing in Europe. In addition, this project will evaluate the performance of various rapid diagnostic tests (RDTs) for SARS-CoV-2, taking into account the above-determined immune system characteristics. In addition, the investigators will evaluate the RDTs for use in the screening of infected patients who are asymptomatic, in particular in health-care settings, as well as for monitoring recovery or clearance of virus shedding for use in resource-constrained setting. Such comparative studies will help identify immune factors that could play a role in attenuating the disrupted immune responses caused by SARS-CoV-2 infection and thus contribute to the design and development of effective diagnostic, therapeutic or vaccine.

The pathogenesis of severe COVID-19 is related to hyper-inflammation. However, COVID-19 symptomatology in SSA appears significantly less serious than in industrialized world. We postulate that individuals residing in SSA and co-infected with intestinal parasites down regulate immune to SARS-CoV-2 and mute COVID-19 severity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical case-definition confirmed by RT-PCR.

Exclusion Criteria:

* Recent history of COVID-19
* Not capable of understanding or complying with the study protocol
* Anticipated transfer to another hospital which is not a study site within 72 hours
* Refusal to consent and participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients suspected of having SARS-CoV-2 infection and admitted to Covid-19 isolation and treatment centers.
Sampling Method: Non-Probability Sample
Enrollment: 838 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients identified as Covid-19 by and monitoring virus clearance with COVID-19 using algorithm of RDTs. | Up to 30 days after onset of infection
  RT-PCR confirmed Covid-19 patients identified by rapid antibody- and antigen-based assays
Proportion of non-Covid-19 cases identified as negative by antibody assay | Up to 30 days after onset of infection other than SARS-CoV-2
  Healthy controls on samples collected pre-Covid-19 pandemic period tested by rapid antibody-based assays

OTHER OUTCOMES:
Proportion of Ethiopian vs. European COVID-19 patients with predominant Th1 type immune responses. | Up to 30 days after onset of infection
  Different immune biomarkers measured in Covid-19 patients presenting with different disease severity stage/spectrum
Proportion of severe COVID-19 patients with or without parasite co-infection | Up to 45 days after onset of infection/during hospitalization)
  Stool exam undertaken among COVID-19 patients presenting with different clinical status at time of admission or isolation
Proportion of patients with SARS-CoV-2 neutralizing antibody titer | Up to 45 days of follow-up after symptom onset
  Measurement of neutralizing antibody titers

CONTACTS AND LOCATIONS:
Overall Officials: Dawit Wolday, MD, PhD, Principal Investigator — Mekelle University
Locations (1):
- Mekelle University College of Health Sciences, Mek'ele, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
Data available upon request and assessment by Ethics Review approvals
Time Frame: Open
Access Criteria: For secondary data analysis, systematic reviews and meta-analysis

REFERENCES:
- [Background] Gebrecherkos T, Challa F, Tasew G, Gessesse Z, Kiros Y, Gebreegziabxier A, Abdulkader M, Desta AA, Atsbaha AH, Tollera G, Abrahim S, Urban BC, Schallig H, Rinke de Wit T, Wolday D. Prognostic Value of C-Reactive Protein in SARS-CoV-2 Infection: A Simplified Biomarker of COVID-19 Severity in Northern Ethiopia. Infect Drug Resist. 2023 May 16;16:3019-3028. doi: 10.2147/IDR.S410053. eCollection 2023. PMID 37215303
- [Result] Gebrecherkos T, Kiros YK, Challa F, Abdella S, Gebreegzabher A, Leta D, Desta A, Hailu A, Tasew G, Abdulkader M, Tessema M, Tollera G, Kifle T, Arefaine ZG, Schallig HH, Adams ER, Urban BC, de Wit TFR, Wolday D. Longitudinal profile of antibody response to SARS-CoV-2 in patients with COVID-19 in a setting from Sub-Saharan Africa: A prospective longitudinal study. PLoS One. 2022 Mar 23;17(3):e0263627. doi: 10.1371/journal.pone.0263627. eCollection 2022. PMID 35320286
- [Result] Wolday D, Gebrecherkos T, Arefaine ZG, Kiros YK, Gebreegzabher A, Tasew G, Abdulkader M, Abraha HE, Desta AA, Hailu A, Tollera G, Abdella S, Tesema M, Abate E, Endarge KL, Hundie TG, Miteku FK, Urban BC, Schallig HHDF, Harris VC, de Wit TFR. Effect of co-infection with intestinal parasites on COVID-19 severity: A prospective observational cohort study. EClinicalMedicine. 2021 Sep;39:101054. doi: 10.1016/j.eclinm.2021.101054. Epub 2021 Jul 31. PMID 34368662
- [Result] Wolday D, Tasew G, Amogne W, Urban B, Schallig HD, Harris V, Rinke de Wit TF. Interrogating the Impact of Intestinal Parasite-Microbiome on Pathogenesis of COVID-19 in Sub-Saharan Africa. Front Microbiol. 2021 Apr 16;12:614522. doi: 10.3389/fmicb.2021.614522. eCollection 2021. No abstract available. PMID 33935986
- [Result] Abraha HE, Gessesse Z, Gebrecherkos T, Kebede Y, Weldegiargis AW, Tequare MH, Welderufael AL, Zenebe D, Gebremariam AG, Dawit TC, Gebremedhin DW, de Wit TR, Wolday D. Clinical features and risk factors associated with morbidity and mortality among patients with COVID-19 in northern Ethiopia. Int J Infect Dis. 2021 Apr;105:776-783. doi: 10.1016/j.ijid.2021.03.037. Epub 2021 Mar 16. PMID 33741488